CLINICAL TRIAL: NCT04739215
Title: Effects of Sodium-Glucose Cotransporter 2 Inhibition on the Mechanisms of Cardiac Damage in the Diabetic Patient With Heart Failure With Preserved Ejection Fraction
Brief Title: Effects of SGLT2 Inhibition on the Mechanisms of Cardiac Damage in the Diabetic Patient With HFpEF
Acronym: CARDIA-STIFF
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital General Universitario Gregorio Marañon (Other)
Collaborators: University of Navarra (Other); Instituto de Salud Carlos III (Other Government); Fundación para la Investigación Biomédica del Hospital Gregorio Maranon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FIBHGM-CARDIA-STIFF; 2019-002046-20 (EudraCT Number)
Record Dates: First submitted 2021-01-15; First posted 2021-02-04 (Actual); Last update posted 2021-02-04 (Actual); Status verified 2021-02

CONDITIONS: Diabetes Mellitus, Type 2; Heart Failure With Preserved Ejection Fraction
Keywords: Diabetes mellitus; Heart Failure
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus; Heart Failure | interventions — dapagliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Clinical Trial: Experimental Arm (Experimental): Patients with heart failure with preserved ejection fraction and type 2 diabetes mellitus treated with Dapagliflozin (Forxiga) 10 mg, one capsule per day orally.
  Interventions: Drug: Dapagliflozin 10 MG [Farxiga]
- Clinical Trial: Placebo Arm (Placebo Comparator): Patients with heart failure with preserved ejection fraction and type 2 diabetes mellitus treated with Placebo in a similar pattern.
  Interventions: Drug: Placebo
- Descriptive Study (No Intervention): Patients with heart failure with preserved ejection fraction but with no type 2 diabetes mellitus (n=10).

INTERVENTIONS:
Drug: Dapagliflozin 10 MG [Farxiga] — Dapagliflozin 10 mg / day oral
  Arms: Clinical Trial: Experimental Arm
Drug: Placebo — One Placebo capsule daily oral
  Arms: Clinical Trial: Placebo Arm

SUMMARY:
The main aim of this study is to identify the underlying mechanisms of Sodium-glucose co-transporter-2 (SGLT2) inhibitors which are associated to better outcomes in patients with Diabetes mellitus type 2 and Heart Failure with preserved Ejection Fraction.

DETAILED DESCRIPTION:
Double design study including a clinical trial and a nested case-control study.

A) Experimental study (clinical trial): Phase IV, prospective, randomized, double-blind placebo-controlled with 12 months follow-up. Inclusion criteria are: 1) diagnosis of DM2, 2) HF with preserved EF with a hospital admission in the previous 6 months with demonstration of diastolic dysfunction. 3) Stable clinical situation at inclusion. 4) Clinical indication of cardiac catheterization.

Patients will be randomized 1:1 to received Dapagliflozin 10 mg/day or placebo. The main objective is to compare the impact of the drug on LV diastolic properties at the peak of effort and in levels of plasma deposit and cross-linking biomarkers of type I collagen between the two treatment groups at baseline and after 12 months.

52 patients will be recruited.

B) Descriptive study: Nested case-control study, considering patients from the experimental study as cases and 10 additional patients with HF with preserved EF but no type 2 DM as controls. The main aim will be compare the histological, molecular, biochemical and biomechanical features of the HFpEF patients with and without DM2.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of DM2 based on the established criteria: HbA1c ≥ 6.5% (48 mmol / mol) and fasting plasma glucose ≥ 7.0 mmol / L (≥126 mg / dL) or 2-h after overload ≥ 11.1 mmol / L ( ≥ 200 mg / dL).
* LVEF ≥ 50%.
* Diagnosis of ICFEP according to clinical criteria, with a hospital admission in the previous 6 months with demonstration of diastolic dysfunction according to the echocardiographic criteria.
* Stable clinical situation (> 1 month after hospitalization due to IC decompensation).
* Clinical indication of cardiac catheterization.
* Signature of informed consent.

Exclusion Criteria:

* Previous treatment with iSGLT2.
* Significant coronary disease.
* Aortic or mitral valve disease ≥ moderate (grades 3 or 4/4 for valve regurgitations)
* Contraindications for dapagliflozin treatment according to the data sheet (hereditary galactose intolerance, Lapp lactase insufficiency or glucose-galactose malabsorption, moderate-severe renal failure -CrCl <60 ml / min or eGFR <60 ml / min / 1 , 73 m2-, severe hepatic insufficiency).

The inclusion/exclusion criteria for Descriptive Study will be the same as previously described without the diagnosis of DM2.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2021-01-15 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Functional Main Objective: Impact of iSGLT2 on LV diastolic properties in terms of the change in LV stiffness constant (S+) at the peak of exercise. | Baseline vs 12 months
  Intrinsic diastolic properties will be analyzed by dynamic pressure-volume loop catheterization.
Main Structural Objective: Changes in serum levels of procollagen type I C-terminal propertied (PICP, ng/mL) | Baseline vs 12 months
  We will measure the changes in serum levels of procollagen type I C-terminal propertied (PICP, ng/mL), a validated biomarker of collagen type I deposition

SECONDARY OUTCOMES:
Changes in LV stiffness constants (S+ and S-). | Baseline vs 12 months
  LV stiffness constants will be obtained from invasive pressure-volume data analysis.
Changes in the slope, Emax, of the end-systolic pressure-volume relationship | Baseline vs 12 months
  Emax will be obtained from invasive pressure-volume data analysis.
Impact of iSGLT2 on myocardial remodeling. | Baseline vs 12 months
  Reverse cardiac remodeling will be studied by cardiac magnetic resonance (CMR). CMR studies will be performed on 1.5 T scanners and will include short-axis cine steady-state free-precession images from base to apex, and standard long axis views for the analysis of mass, volume and ventricular function.
  CMR study will require the administration of a gadolinium contrast medium to study myocardial fibrosis, unless contraindicated.
Correlation of myocardial remodeling patterns with the intrinsic diastolic properties of chamber VI with systolic function. | Baseline vs 12 months
  Results from the pressure-volume analysis and CMR will be assess in common in order to search for association.
Relative contribution of the intrinsic diastolic properties of the LV and the flow patterns on filling pressures and their modulation under treatment with iSGLT2. | Baseline vs 12 months
  Intraventricular flow patterns will be studied by Doppler echocardiography and phase contrast CMR, considering vorticity and blood transport parameters.
Changes in serum levels of collagen type I C-terminal telopeptide to matrix metalloproteinase ratio (CITP:MMP-1) | Baseline vs 12 months
  We will measure the changes in serum levels of collagen type I C-terminal telopeptide to matrix metalloproteinase ratio (CITP:MMP-1), biomarker of the degree of collagen type cross-linking.
Changes in N-terminal pro brain natriuretic peptide (pg/mL) | Baseline vs 12 months
  We will measure the changes in N-terminal pro brain natriuretic peptide (pg/mL)
Changes in high sensitivity troponin T (pg/mL) | Baseline vs 12 months
  We will measure the changes in high sensitivity troponin T (pg/mL)

CONTACTS AND LOCATIONS:
Overall Officials: Javier Bermejo Thomas, MD, PhD, Principal Investigator — Hospital General Universitario Gregorio Marañón
Locations (1):
- Hospital General Universitario Gregorio Maranon, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Kasner M, Westermann D, Lopez B, Gaub R, Escher F, Kuhl U, Schultheiss HP, Tschope C. Diastolic tissue Doppler indexes correlate with the degree of collagen expression and cross-linking in heart failure and normal ejection fraction. J Am Coll Cardiol. 2011 Feb 22;57(8):977-85. doi: 10.1016/j.jacc.2010.10.024. PMID 21329845
- [Result] Zinman B, Wanner C, Lachin JM, Fitchett D, Bluhmki E, Hantel S, Mattheus M, Devins T, Johansen OE, Woerle HJ, Broedl UC, Inzucchi SE; EMPA-REG OUTCOME Investigators. Empagliflozin, Cardiovascular Outcomes, and Mortality in Type 2 Diabetes. N Engl J Med. 2015 Nov 26;373(22):2117-28. doi: 10.1056/NEJMoa1504720. Epub 2015 Sep 17. PMID 26378978
- [Result] Perez Del Villar C, Savvatis K, Lopez B, Kasner M, Martinez-Legazpi P, Yotti R, Gonzalez A, Diez J, Fernandez-Aviles F, Tschope C, Bermejo J. Impact of acute hypertension transients on diastolic function in patients with heart failure with preserved ejection fraction. Cardiovasc Res. 2017 Jul 1;113(8):906-914. doi: 10.1093/cvr/cvx047. PMID 28402411
- [Result] Bermejo J, Yotti R, Perez del Villar C, del Alamo JC, Rodriguez-Perez D, Martinez-Legazpi P, Benito Y, Antoranz JC, Desco MM, Gonzalez-Mansilla A, Barrio A, Elizaga J, Fernandez-Aviles F. Diastolic chamber properties of the left ventricle assessed by global fitting of pressure-volume data: improving the gold standard of diastolic function. J Appl Physiol (1985). 2013 Aug 15;115(4):556-68. doi: 10.1152/japplphysiol.00363.2013. Epub 2013 Jun 6. PMID 23743396